CLINICAL TRIAL: NCT02734953
Title: Effects of iNO on Invasively Derived Pulmonary Vascular Parameters in Patients With Pulmonary Arterial Hypertension
Brief Title: Effect of iNO on Invasively Derived Pulmonary Pressures in Patients With PAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Raymond Benza, Physician, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC6167
Record Dates: First submitted 2016-03-26; First posted 2016-04-12 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Inhaled nitric oxide; Exercise; 6 minute walk test; CardioMems
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Motor Activity | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Determination of non-invasive pulmonary pressures by CardioMems device interrogation pre- and post-administration of inhaled nitric oxide at 0.075 mg/kg IBW/hr
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Ambulatory inhaled nitric oxide delivery system and 6 minute walk distance test
  Other Names: iNOPulse DS

SUMMARY:
Pulmonary hypertension is characterized by an increase in the pressures in the blood supply to the lungs greater than a mean pressure of 25mmHg and a concomitant increase in overall pulmonary vascular resistance (PVR). In patients who have remodeling of their pulmonary vasculature, PVR will increase with exercise instead of decreasing as it would in normal patients. Based on published evidence, the investigators intend to investigate the effects of inhaled nitric oxide (iNO) on patients undergoing standard exercise techniques who have separately and previously had an implanted pulmonary artery monitoring device (CardioMems by St Jude Medical, Inc.) placed.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18 to 80 years with a diagnosis of pulmonary arterial hypertension (WHO Group I pulmonary hypertension).
* Must be able to read and understand English and consent for themselves
* Previously implanted CardioMems continuous PA pressure
* Ambulatory and able to complete 6MWD test.

Exclusion Criteria:

* Pregnant or lactating females; negative pregnancy test as confirmed by evaluation of data from pre-enrolled Risk Evaluation and Mitigation Strategies (REMS) program.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Benza, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
With sponsor to provide statistical analysis

REFERENCES:
- [Background] Frantz RP, Benza RL, Kjellstrom B, Bourge RC, Barst RJ, Bennett TD, McGoon MD. Continuous hemodynamic monitoring in patients with pulmonary arterial hypertension. J Heart Lung Transplant. 2008 Jul;27(7):780-8. doi: 10.1016/j.healun.2008.04.009. Epub 2008 Jun 2. PMID 18582809
- [Background] Hasuda T, Satoh T, Shimouchi A, Sakamaki F, Kyotani S, Matsumoto T, Goto Y, Nakanishi N. Improvement in exercise capacity with nitric oxide inhalation in patients with precapillary pulmonary hypertension. Circulation. 2000 May 2;101(17):2066-70. doi: 10.1161/01.cir.101.17.2066. PMID 10790348
- [Background] Kjellstrom B, Frantz RP, Benza RL, Bennett T, Bourge RC, McGoon MD. Hemodynamic ranges during daily activities and exercise testing in patients with pulmonary arterial hypertension. J Card Fail. 2014 Jul;20(7):485-91. doi: 10.1016/j.cardfail.2014.04.019. Epub 2014 May 9. PMID 24816520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: June 1-25, 2016 Recruitment Location: medical clinic
Pre-assignment Details: All enrolled participants were included,
Period: Overall Study
Arm/Group | Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Difference in Ambulatory 6 Minute Walk Distance (6MWD) Pulmonary Artery (PA) Pressures (Systolic, Diastolic, Mean) Between the Post-intervention (iNO+) and Pre-intervention (iNO-) Condition as Measured by the CardioMems Device
Description: Difference between baseline (t=0) and post-intervention (t=2h)
Time Frame: 2 hours
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Intervention
Number analyzed (Participants) | 10
mmHg
  PA pressure systolic | -4.86 [-22.96 to 9.31]
  PA pressure diastolic | -2.40 [-10.54 to 7.8]
  PA pressure mean | -3.45 [-14.97 to 9.85]

2. Secondary Outcome: Change in CardioMems Cardiac Output
Description: Difference between baseline (t=0) and post-intervention (t=2h)
Time Frame: 2 hours
Measure: Mean (Full Range); unit: L/min
Arm/Group | Intervention
Number analyzed (Participants) | 10
L/min | 0.76 [-1.34 to 5.26]

3. Secondary Outcome: Change in 6 Minute Walk Distance (6MWD)
Description: Difference (in distance walked between 2 set points over 6 minutes) at baseline (t=0) to post-intervention (t=2h).
Time Frame: 2 hours
Measure: Mean (Full Range); unit: m
Arm/Group | Intervention
Number analyzed (Participants) | 10
m | 12.6 [-16 to 55]

4. Secondary Outcome: Change in O2 Saturations
Time Frame: 2 hours
Measure: Mean (Full Range); unit: % O2 Sat
Arm/Group | Intervention
Number analyzed (Participants) | 10
% O2 Sat | -1 [-3 to 2]

5. Secondary Outcome: Change in Modified Borg Dyspnea Scale
Description: The Modified Borg Dyspnea scale measures patient's subjective analysis of dyspnea from 0 ("nothing at all") to 10 ("maximal") during the 6MWD test with the highest value recorded and difference calculated between baseline (t=0) and post-intervention (t=2h).
Time Frame: 2 hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
units on a scale | -0.4 [-2 to 1]

6. Secondary Outcome: Change in O2 Requirements
Description: Number of patients that required more or less oxygen by nasal prongs during the course of the study.
Time Frame: 2 hours
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 10
participants | 0

7. Secondary Outcome: Change in Mean Arterial Pressure
Description: Difference between baseline (t=0) and post-intervention (t=2h).
Time Frame: 2 hours
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Intervention
Number analyzed (Participants) | 10
mmHg | -7 [-17 to -1]

8. Secondary Outcome: Change in Heart Rate
Description: Difference between baseline (t=0) and post-intervention (t=2h)
Time Frame: 2 hours
Measure: Mean (Full Range); unit: bpm
Arm/Group | Intervention
Number analyzed (Participants) | 10
bpm | 4 [-25 to 45]

9. Secondary Outcome: Change in Rate Pressure Product
Description: Difference between baseline (t=0) and post-intervention (t=2h)
Time Frame: 2 hours
Measure: Mean (Full Range); unit: mmHg*beat/min
Arm/Group | Intervention
Number analyzed (Participants) | 10
mmHg*beat/min | 316 [-3490 to 8900]

10. Secondary Outcome: Change in Right Ventricular (RV) Power
Description: Difference between baseline (t=0) and post-intervention (t=2h)
Time Frame: 2 hours
Measure: Mean (Full Range); unit: J/s
Arm/Group | Intervention
Number analyzed (Participants) | 10
J/s | 0.00685 [-0.150 to 0.241]

11. Secondary Outcome: Change in Stroke Volume
Description: Difference between baseline (t=0) and post-intervention (t=2h)
Time Frame: 2 hours
Measure: Mean (Full Range); unit: mL
Arm/Group | Intervention
Number analyzed (Participants) | 10
mL | 2.97 [-20.8 to 28.0]

12. Secondary Outcome: Change in RV Stroke Work Index
Description: Difference between baseline (t=0) and post-intervention (t=2h)
Time Frame: 2 hours
Measure: Mean (Full Range); unit: g*m/m2
Arm/Group | Intervention
Number analyzed (Participants) | 10
g*m/m2 | -1.80 [-11.6 to 1.53]

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No